CLINICAL TRIAL: NCT01690390
Title: An Open-label, Randomized, Multicenter, Phase II Trial to Evaluate the Safety and Efficacy of Dose Escalation of Icotinib in Advanced or Metastatic NSCLC Patients After 8 Weeks Routine Therapy Evaluated as Stable Disease
Brief Title: Dose Escalation of Icotinib in Advanced Non-small Cell Lung Carcinoma (NSCLC) Patients Evaluated as Stable Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IV-43
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2013-12

CONDITIONS: NSCLC
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib of Routine Dose (Active Comparator): Oral Drug icotinib 125 mg three times per day
  Interventions: Drug: Icotinib of routine dose
- Icotinib of High Dose (Experimental): Oral Drug icotinib 250 mg three times per day
  Interventions: Drug: Icotinib of high dose

INTERVENTIONS:
Drug: Icotinib of routine dose — Icotinib of routine dose: 125 mg is administered orally three times per day.
  Other Names: Icotinib; Comana; BPI-2009
  Arms: Icotinib of Routine Dose
Drug: Icotinib of high dose — Icotinib: 250 mg is administered orally three times per day.
  Other Names: Icotinib; Comana; BPI-2009
  Arms: Icotinib of High Dose

SUMMARY:
The primary purposes of this study are to assess the safety and efficacy of using high doses of the drug Icotinib (Conmana) as a way to treat patients with non-small cell lung cancer that achieve stable disease after 8 weeks routine therapy.

DETAILED DESCRIPTION:
This is a multi-center phase II randomized controlled study to assess the safety and efficacy of using high doses of the drug Icotinib (Conmana) as a way to treat patients with non-small cell lung cancer that achieve stable disease after 8 weeks routine therapy by PFS, as well as OS and DCR. The adverse events and adverse reaction are evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV lung cancer(exclude patients confirmed by sputum cytology)
* No previous targeted treatment such as gefitinib, erlotinib.
* With a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) at least according to RECIST Criteria
* WHO performance status(PS)<= 2
* N>=1.5×109/L, Plt>=1.0×109/L,Hb>=10g/dL;AST&ALT should <3ULN(without liver metastasis) or <5ULN(with liver metastasis).TBIL<=1.5ULN.
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Allergic to icotinib
* Patients with metastatic brain tumors with symptoms.
* Experience of Anti-EGFR(the epidermal growth factor receptor) Monoclonal Antibody or small molecular compounds therapy such as gefitinib, erlotinib or Cetuximab.
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival | 15 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.
Transformation rate from stable disease to complete response or partial response | 6 weeks
  Number of participants with an stable disease previously achieve complete response or partial response after dose escalation. Either complete response (CR) or partial response (PR) will be evaluated by RECIST, confirmed at least 28 days following the date of the initial response.
Incidence rate of adverse events | 40 months
  Number of patients with a adverse event, identified according to the Common Toxicity Criteria (CTC) in evaluable-for-safety population, which included all patients who received at least 1 dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yi Ping, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (17):
- China (17):
  - Fujian Hospital for Chest Tumors & Tuberculosis Diseases, Fuzhou, Fujian
  - Fujian Provincal Hospital, Fuzhou, Fujian
  - Fujian Provincal Cancer Hospital, Fuzhou, Fujian
  - The second hospital of Xiamen City, Xiamen, Fujian
  - Hunan Provincal Cancer Hospital, Changsha, Hunan
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Traditional Chinese Medical Hospital, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Yinzhou People's Hospital, Ningbo, Zhejiang
  - Ningbo Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang